CLINICAL TRIAL: NCT03883178
Title: New Endoscopic Minimal Invasive Approach for Pudendal Nerve and Inferior Cluneal Nerve Neurolysis: a Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katleen JOTTARD (Other)
Responsible Party: Sponsor-Investigator, Katleen JOTTARD, Deputy Chief of Clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUB-neurolysis
Record Dates: First submitted 2019-03-15; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Pudendopathie; Clunealgie

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurolysis (Experimental)
  Interventions: Procedure: Minimal-invasive endoscopic transgluteal approach

INTERVENTIONS:
Procedure: Minimal-invasive endoscopic transgluteal approach — Every patient, suffering from a pudendopathie or clunealgie, conform the Nantes criteria, and who are candidates for a surgical treatment through the transgluteal open approach, will be asked their permission to perform the procedure through a minimal-invasive endoscopic transgluteal approach.

SUMMARY:
Pudendal nerve and cluneal nerve entrapment can cause a neuropathic pain syndrome in one, many or all of the sensitive areas innervated by this nerve. In literature, several techniques for the liberation of the pudendal nerve have been described. Here, transvaginal, transperineal and abdominal laparoscopic approaches have been proposed, but none of the latter were able to visualize the entire course of the nerve or allowed to explore the main, currently identified sites of entrapment. Although there have been reports and series of case reports on different surgical approaches, until now, the transgluteal approach is the only one which is validated by a prospective randomized study comparing the medical treatment to these surgical approach.

The investigators already performed a study to describe for the first time a new endoscopic minimal invasive technique using a transgluteal approach which permits to visualize all the nerve structures of the gluteal region. They performed an anatomic description of the region reachable with this minimally invasive approach, and described the anatomic landmarks for the visualization of the pudendal and cluneal nerve and their neurolysis.

In this study, the investigators would like to put in clinical practice this minimal invasive approach for pudendal and cluneal neurolysis. They will perform this endoscopic approach, on patients suffering from pudendalgie or/and clunealgie, who are programmed for a surgical intervention by transgluteal approach.

The investigators would like to test the feasibility of the transgluteal trocar positioning and if necessary, optimize this first important step. Secondly, they will put in practice the step-by-step surgical approach that they have worked out during their cadaver study. Finally, they will perform the entire neurolysis and nerve transposition under endoscopic control.

ELIGIBILITY:
Inclusion Criteria:

Patients suffering from pudendalgie and/ or clunealgie, according to the 5 Nantes criteria and who are candidates for transgluteal surgical treatment.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
score on the SF-36 questionnaire | Change from baseline at 3 months after surgery
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. It covers several health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.The recommended scoring system for the SF-36 is a weighted Likert system for each item. The items in the subscales are summed to obtain a summary score for each subscale or dimension. Each of the 8 summary scores is linearly transformed on a scale of 0 (negative to health) to 100 (positive for health).
Pain intensity according to EVA scale | Change from baseline at 3 months after surgery
  Linear scale raging from 0 (no pain) to 10 (maximal pain).
Pain intensity according to EVA scale | Change from baseline at 6 months after surgery
  Linear scale raging from 0 (no pain) to 10 (maximal pain).
Surgery duration | 24 hours
  Surgery duration
Adverse events during surgery | 24 hours
  Exhaustive list of the adverse events occuring during surgery
Adverse events after surgery | 48 hours
  Exhaustive list of the adverse events occuring after surgery.
Conversion rate | 24 hours
  Rate of conversions from the minimal-invasive endoscopic transgluteal approach to the open transgluteal approach during the surgery.
Number of trocars used during surgery | 24 hours
  Number of 5 mm trocars used in transgluteal position during the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Katleen Jottard, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Labat JJ, Riant T, Robert R, Amarenco G, Lefaucheur JP, Rigaud J. Diagnostic criteria for pudendal neuralgia by pudendal nerve entrapment (Nantes criteria). Neurourol Urodyn. 2008;27(4):306-10. doi: 10.1002/nau.20505. PMID 17828787
- [Background] Ploteau S, Salaud C, Hamel A, Robert R. Entrapment of the posterior femoral cutaneous nerve and its inferior cluneal branches: anatomical basis of surgery for inferior cluneal neuralgia. Surg Radiol Anat. 2017 Aug;39(8):859-863. doi: 10.1007/s00276-017-1825-z. Epub 2017 Feb 24. PMID 28236130
- [Background] Beco J, Climov D, Bex M. Pudendal nerve decompression in perineology: a case series. BMC Surg. 2004 Oct 30;4:15. doi: 10.1186/1471-2482-4-15. PMID 15516268
- [Background] Erdogru T, Avci E, Akand M. Laparoscopic pudendal nerve decompression and transposition combined with omental flap protection of the nerve (Istanbul technique): technical description and feasibility analysis. Surg Endosc. 2014 Mar;28(3):925-32. doi: 10.1007/s00464-013-3248-1. Epub 2013 Oct 23. PMID 24149853
- [Background] Konschake M, Brenner E, Moriggl B, Hormann R, Bauer S, Foditsch E, Janetschek G, Kunzel KH, Sievert KD, Zimmermann R. New laparoscopic approach to the pudendal nerve for neuromodulation based on an anatomic study. Neurourol Urodyn. 2017 Apr;36(4):1069-1075. doi: 10.1002/nau.23090. Epub 2016 Aug 4. PMID 27490402
- [Background] Robert R, Labat JJ, Bensignor M, Glemain P, Deschamps C, Raoul S, Hamel O. Decompression and transposition of the pudendal nerve in pudendal neuralgia: a randomized controlled trial and long-term evaluation. Eur Urol. 2005 Mar;47(3):403-8. doi: 10.1016/j.eururo.2004.09.003. PMID 15716208
- [Derived] Jottard K, Bruyninx L, Bonnet P, De Wachter S. Endoscopic trans gluteal minimal-invasive approach for nerve liberation (ENTRAMI technique) in case of pudendal and/or cluneal neuralgia by entrapment: One-year follow-up. Neurourol Urodyn. 2020 Sep;39(7):2003-2007. doi: 10.1002/nau.24462. Epub 2020 Jul 17. PMID 32678485
- [Derived] Jottard K, Bruyninx L, Bonnet P, De Wachter S. A minimally invasive, endoscopic transgluteal procedure for pudendal nerve and inferior cluneal nerve neurolysis in case of entrapment: 3- and 6-month results. The ENTRAMI technique for neurolysis. Int J Colorectal Dis. 2020 Feb;35(2):361-364. doi: 10.1007/s00384-019-03480-2. Epub 2019 Dec 11. PMID 31828369